CLINICAL TRIAL: NCT04866173
Title: Effects of Contact to a Dog During Standardised Stressful Situations
Brief Title: Effects of Contact to Dogs During Stressful Situations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ANIMAL CONTACT2; 128534 (Other Grant/Funding Number: TrygFonden)
Record Dates: First submitted 2021-04-14; First posted 2021-04-29 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-04

CONDITIONS: Physiological Stress Responses to Standardises Stress Situations; Psychological Responses to Standardised Stress Situations; Behavioural Responses to Standardised Stress Situations
Keywords: Human-animal contact; Non-invasive measure; Animal-assisted contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dog (Experimental): Being subjected to two standardised stress situations with a dog and its handler present
  Interventions: Other: Dog
- No Dog (Experimental): Being subjected to two standardised stress situations without a dog present, but in the presence of a person (dog handler)
  Interventions: Other: No Dog

INTERVENTIONS:
Other: Dog — Subjection to standardised stress situations in the presence of a dog and a person
  Arms: Dog
Other: No Dog — Subjection to standardised stress situations in the presence of a person
  Arms: No Dog

SUMMARY:
The investigators will conduct an experimental study comparing responses of healthy participants in two test situations where they are subjected to mild stress. The study design is a randomised controlled crossover design nested within two groups - one with a dog present and another without a dog present. The participants will be randomly allocated to two groups (with dog and without dog) and the participants will receive both test situations on the same day. During the two test situations the participants will be subjected to a classical stress test , and exposed to tolerable pain, as well as periods with relaxation.

DETAILED DESCRIPTION:
The study design is a randomised controlled crossover design, nested within two groups - one with a dog present (Dog) and another without a dog present (No Dog). Both groups will be subjected to a classical stress test - the Maastricht Acute Stress Test (MAST) and a pain test with periods of relaxation in between. The participants will be subjected to both test situations on the same day and in the same order.

On the test day, background information and baseline measures (baseline period, duration: 40 minutes) will be collected, whereafter the participants rest for 30 minutes (pre-intervention rest period). After this the participants are subjected to the two test situations, pain test (60 minutes, including calibration and two separate tests sessions) and MAST (15 minutes, including 5 min introduction) with 30 minutes of relaxation in between and a 40 min post-rest period The participants' interaction with the dog is recorded using quantitative behaviour sampling using predefined behavioural categories.

Most physiological and all behavioural measures are recorded continuously throughout test situations and relaxation, in order to be able to study the response to the stress situations and recovery, and the response to contact with dog, and to psychological responses. Some physiological measures obtained before and after each test situation.

Below the exact time schedule of the test day is shown and these times will be refered to when the outcome measures are described. The "Baseline period" (40 minutes) and the last 10 minutes where the equipment for physiological measures is removed is not included in the duration of the test period (174 minutes). All times are given in minutes.

Baseline period (40 minutes - not part of total test period)

* Pre-intervention period (start t = 0; end t = 30)
* Calibration for pain test (start t = 30, end t = 35)
* Rest period 1 (start t = 35, end t = 47)
* Pain test 1 (start t = 47, end t = 52)
* Post-pain test 1 (start t = 52, end, t= 62)
* Rest period 2 (start t = 62, end t = 74)
* Pain test 2 (start t = 74, end t = 79)
* Post-pain test 2 (start t = 79, end t = 89)
* Rest period 3 (start t = 89, end t = 119)
* MAST test (incl. introduction (start t = 119, end t = 134)
* Rest period 4 (start t = 134, end t = 174)

ELIGIBILITY:
Inclusion Criteria:

* Normal cognitive functioning and physical movement
* Ability to speak and read Danish

Exclusion Criteria:

* Known medical, psychiatric or neurological disease
* Use of psychotropic medications
* Frequent use of pain medication
* Use of illegal psychotropic drugs
* Known allergies to dogs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-10-17 (Actual)

PRIMARY OUTCOMES:
Physiological measure, heart rate | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  The test person wears self-adhesive electrodes and the heart rate is measured non-invasively
Physiological measure, systolic and diastolic blood pressure | Measured at the end of the 30 minute pre-intervention period (t=30 minutes)]
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff.
Physiological measure, systolic and diastolic blood pressure | Measured at the end of Rest Period 1 (t=47 minutes)]
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff.
Physiological measure, systolic and diastolic blood pressure | Measured after Pain test 1 (t=52 minutes)]
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff.
Physiological measure, systolic and diastolic blood pressure | Measured at the end of Rest period 2 (t=74 minutes)]
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff.
Physiological measure, systolic and diastolic blood pressure | Measured after Pain test 2 (t=79 minutes)]
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff.
Physiological measure, systolic and diastolic blood pressure | Measured at the end of Rest period 3 (t=119 minutes)]
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff.
Physiological measure, systolic and diastolic blood pressure | Measured after MAST test (t=134 minutes)]
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Physiological measure, systolic and diastolic blood pressure | Measured after Rest period 4 (t=174 minutes)]
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff.
Physiological measure, heart rate variability | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  Heart rate variability is calculated from heart rate data.
Galvanic skin response | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  The test person is fitted with electrodes on two fingers and galvanic skin response is measured non-invasively.
Salivary cortisol | Measured at the end of the 30 minute pre-intervention period (t=30 minutes)]
  Saliva is obtained from the test subject with a cotton swab which is chewed for one minute.
Salivary cortisol | Measured at the end of Rest Period 1 (t=47 minutes)]
  Saliva is obtained from the test subject with a cotton swab which is chewed for one minute
Salivary cortisol | Measured after Post-pain test 1 (t=62 minutes)]
  Saliva is obtained from the test subject with a cotton swab which is chewed for one minute
Salivary cortisol | Measured at the end of Rest period 2 (t=74 minutes)]
  Saliva is obtained from the test subject with a cotton swab which is chewed for one minute
Salivary cortisol | Measured after Post-pain test 2 (t=89 minutes)]
  Saliva is obtained from the test subject with a cotton swab which is chewed for one minute
Salivary cortisol | Measured at the end of Rest period 3 (t=119 minutes)]
  Saliva is obtained from the test subject with a cotton swab which is chewed for one minute
Salivary cortisol | Measured after MAST test (t=134 minutes)]
  Saliva is obtained from the test subject with a cotton swab which is chewed for one minute
Salivary cortisol | Measured 5 minutes after MAST test (t=139 minutes)]
  Saliva is obtained from the test subject with a cotton swab which is chewed for one minute
Salivary cortisol | Measured 10 minutes after MAST test (t=144 minutes)]
  Saliva is obtained from the test subject with a cotton swab which is chewed for one minute
Salivary cortisol | Measured 20 minutes after MAST test (t=154 minutes)]
  Saliva is obtained from the test subject with a cotton swab which is chewed for one minute
Salivary cortisol | Measured 30 minutes after MAST test (t=164 minutes)]
  Saliva is obtained from the test subject with a cotton swab which is chewed for one minute
Salivary cortisol | Measured 40 minutes after MAST test (t=174 minutes)]
  Saliva is obtained from the test subject with a cotton swab which is chewed for one minute
Visual analogue scales measuring expected psychological and physiological effects of the test day including, including the two test situation and the rest periods | Baseline: Measured at onset of the 30 minute pre-intervention period (t=0 minutes)]
  Test persons fill in a visual analogue scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring expected psychological and physiological effects of the two test situations | : Measured immediately preceding Pain test 1 (t=47 minutes]
  Test persons fill in a visual analogue scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring expected psychological and physiological effects of the two test situations | : Measured immediately preceding Pain test 2 (t=74 minutes]
  Test persons fill in a visual analogue scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring expected psychological and physiological effects of the two test situations | : Measured immediately preceding MAST test (t=119 minutes]
  Test persons fill in a visual analogue scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring perceived psychological and physiological effects of each of the two test situations | Measured immediately following Pain test 1(t=52 minutes)
  Test persons fill in a visual analogue scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring perceived psychological and physiological effects of each of the two test situations | Measured immediately following Pain test 2 (t=79 minutes)
  Test persons fill in a visual analogue scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring perceived psychological and physiological effects of each of the two test situations | Measured immediately following MAST test 1 (t=134 minutes)
  Test persons fill in a visual analogue scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring perceived psychological and physiological effects of of the test day including the test situations and rest period | Measured immediately after Rest period 4 (t=174 minutes)
  Test persons fill in a visual analogue scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
The State-Trait Anxiety Inventory (STAI) | Baseline: Measured at onset of the 30 minute pre-intervention period preceding the first test situation (t=0 minutes)]
  State anxiety is measured with the STAI-scale (minimum score= 20, maximum score= 80, and a lower score indicates a high anxiety level)
The State-Trait Anxiety Inventory (STAI) | Measured immediately following Pain test 1 (t= 52 minutes)
  State anxiety is measured with the STAI-scale (minimum score= 20, maximum score= 80, and a lower score indicates a high anxiety level)
The State-Trait Anxiety Inventory (STAI) | Measured immediately following Pain test 2 (t= 79 minutes)
  State anxiety is measured with the STAI-scale (minimum score= 20, maximum score= 80, and a lower score indicates a high anxiety level)
The State-Trait Anxiety Inventory (STAI) | Measured immediately following MAST test 1 (t=134 minutes)
  State anxiety is measured with the STAI-scale (minimum score= 20, maximum score= 80, and a lower score indicates a high anxiety level)
The State-Trait Anxiety Inventory (STAI) | Measured immediately after Rest period 4 (t=174 minutes)
  State anxiety is measured with the STAI-scale (minimum score= 20, maximum score= 80, and a lower score indicates a high anxiety level)
The Positive and Negative Affect Schedule (PANAS) | Baseline: Measured at onset of the 30 minute pre-intervention period preceding the first test situation (t=0 minutes)]
  Positive and negative affect is measured with the PANAS scale, where the person scores whether or not they experience each of 20 emotions on a 5-step scale from "very little /not at all" to "extremely much". The emotions differ in valens.
The Positive and Negative Affect Schedule (PANAS) | Measured immediately following Pain test 1 (t= 52 minutes)
  Positive and negative affect is measured with the PANAS scale, where the person scores whether or not they experience each of 20 emotions on a 5-step scale from "very little /not at all" to "extremely much". The emotions differ in valens.
The Positive and Negative Affect Schedule (PANAS) | Measured immediately following Pain test 2 (t= 79 minutes)
  Positive and negative affect is measured with the PANAS scale, where the person scores whether or not they experience each of 20 emotions on a 5-step scale from "very little /not at all" to "extremely much". The emotions differ in valens.
The Positive and Negative Affect Schedule (PANAS) | Measured immediately following MAST test 1 (t=134 minutes)
  Positive and negative affect is measured with the PANAS scale, where the person scores whether or not they experience each of 20 emotions on a 5-step scale from "very little /not at all" to "extremely much". The emotions differ in valens.
The Positive and Negative Affect Schedule (PANAS) | Measured immediately after Rest period 4 (t=174 minutes)
  Positive and negative affect is measured with the PANAS scale, where the person scores whether or not they experience each of 20 emotions on a 5-step scale from "very little /not at all" to "extremely much". The emotions differ in valens.
Quantitative behavioural measures - frequencies of behavioural elements | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  A video recording of the test persons behaviour is analysed for frequency of sitting.
Quantitative behavioural measures - frequencies of behavioural elements | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  A video recording of the test persons behaviour is analysed for frequency of standing.
Quantitative behavioural measures - frequencies of behavioural elements | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  A video recording of the test persons behaviour is analysed for frequency of walking.
Quantitative behavioural measures - frequencies of behavioural elements | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  A video recording of the test persons behaviour is analysed for frequency of touching the dog (being in physical contact with the dog with the hand or another part of the body, only in the arm: Dog)
Quantitative behavioural measures - frequencies of behavioural elements | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  A video recording of the test persons behaviour is analysed for frequency of looking at the dog (having the head turned towards the dog, only in the arm: Dog).
Quantitative behavioural measures - frequencies of behavioural elements | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  A video recording of the test persons behaviour is analysed for frequency of talking to the dog (Only in the arm: Dog).
Quantitative behavioural measures - duration of behavioural elements | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  A video recording of the test persons behaviour is analysed for the duration (seconds) of sitting.
Quantitative behavioural measures - duration of behavioural elements | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  A video recording of the test persons behaviour is analysed for the duration (seconds) of standing.
Quantitative behavioural measures - duration of behavioural elements | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  A video recording of the test persons behaviour is analysed for the duration (seconds) of walking.
Quantitative behavioural measures - duration of behavioural elements | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  A video recording of the test persons behaviour is analysed for the duration (seconds) of touching the dog (being in physical contact with the dog with the hand or another part of the body, only in the arm: Dog).
Quantitative behavioural measures - duration of behavioural elements | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  A video recording of the test persons behaviour is analysed for the duration (seconds) of looking at the dog (having the head turned towards the dog, only in the arm: Dog).
Quantitative behavioural measures - duration of behavioural elements | Measured continuously throughout the total test period of 174 minutes (starting in the pre-intervention period and during the following test situations and all resting periods)]
  A video recording of the test persons behaviour is analysed for the duration (seconds) of talking to the dog (Only in the arm: Dog).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Thodberg, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Tjele, Denmark

IPD SHARING:
Plan to Share IPD: No